CLINICAL TRIAL: NCT05354856
Title: The Effect of Chemoradiotherapy on Gastric Perfusion in Patients With Gastric Cancer.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruiting issues
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, JENS OSTERKAMP, MD, PhD-student, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-20027060
Record Dates: First submitted 2022-02-15; First posted 2022-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Only patients with resectable gastric cancer are included in the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG patient (Experimental): All patients included in the study will be injected with ICG (0.2 mg/kg bodyweight) to assess gastric perfusion.
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — A bolus of ICG (0.2 mg/kg body weight) will be injected intravenously and flushed with 5 mL of saline. Gastric perfusion will subsequently be assessed along specific regions of interest (ROI) with q-ICG (quantitative perfusion assessments with ICG) to obtain baseline perfusion values.

SUMMARY:
A study from our group (Osterkamp et al. in preparation) used ICG to evaluate intraoperative changes in gastric perfusion when reducing the circulating blood volume by blood withdrawal in pigs. We saw a significant reduction in gastric perfusion with decreased blood volume, and this reduction of gastric perfusion was detectable with ICG. As data from a previous trial (PRESET phase 2 Protocol nr: H-15014904) has shown that chemotherapy decreases the circulating red blood cell volume in patients with gastroesophageal cancer, we wish to evaluate if standard care neoadjuvant chemotherapy also influences gastric perfusion. Gastric perfusion will be assessed during a screening laparoscopy (before chemotherapy) and then compared with a second assessment during gastric resection (after chemotherapy). The gastric perfusion will be measured using fluorescence-guided surgery with Indocyanine Green.

Participants will be offered the opportunity to have their blood volume measured during the trial. This is not required in order to take part in the fluorescence angiography part of the study.

DETAILED DESCRIPTION:
Screening Laparoscopy:

As part of the standard care for gastric cancer, all patients undergo a screening laparoscopy before entering neoadjuvant chemotherapy. The procedure is performed to detect overt metastases not detected on the CT/PET-CT scans. First, the patient is placed under a standardized general anesthesia, and the laparoscopic set-up is completed. After anesthesia a peripheral arterial catheter will be placed in order acquire reading of cardia output and stroke volume. The patient will then be fluid optimized using a standardized stroke volume (SV) optimization algorithm. The abdomen is inspected visually for signs of metastatic disease. The small bowel is then manipulated, allowing for visualization of the stomach. A bolus of ICG (0.2 mg/kg body weight) will be injected intravenously and flushed with 5 mL of saline. Gastric perfusion will subsequently be assessed along specific regions of interest (ROI) with q-ICG to obtain baseline perfusion values.

As a substudy, 10 patients will have two measurements with ICG during the screening laparoscopy, one befor eand one after fluid optimization. These patients will receive an ICG dose of 0.1 mg/kg body weight per measurement, totalling 0.2 mg/kg after the two measurements.

Resection of gastric cancer:

The patient is placed under general anesthesia and after the stomach is visualized through surgical incision, a bolus of ICG (0.2 mg/kg body weight) will be injected intravenously and flushed with 5 mL of saline. The ROIs (the same ROIs as described in 3.7.1) will then be assessed with q-ICG. The anesthetic protocol will up to this point match that of the setting during the screening laparoscopy.

Fluorescence angiography:

During the screening laparoscopy, a laparoscope (telescope 30°, 5 mm, Arthrex Danmark A/S) will be connected to a camera system (Synergy, Arthrex Danmark A/S) and a light-source (Synergy Laser Light Source, Arthrex Danmark A/S) will supply the excitatory light and record the ICG angiography. The laparoscope will be fixed in a mechanical holding arm 10 cm from the tissue of interest, ensuring a stable position throughout the experiment.

Measuring of blood volume:

Hemoglobin mass (Hbmass) will be determined using a carbon monoxide (CO) rebreathing technique with a typical error of 1.0 %, as previously described (25). In brief, all individuals will rest for 20 min in the supine position before each measurement. During this time, a catheter will be inserted in an antecubital vein. Thereafter, 2 ml of blood will be sampled and analyzed immediately in triplicates for percentage carboxyhaemoglobin (% HbCO) and [Hb] (ABL800, Radiometer, Denmark). Subsequently, individuals will breathe 100 % O2 for 4 min to flush nitrogen from the airways. Then, a bolus of 1.5 ml kg-1 of 99.997 % chemically pure CO (CO N47, Air Liquide, France) will be administrated into the breathing circuit. Individuals will re-breath this gas mixture for 10 min. An additional 2 ml blood sample will be obtained and analyzed in triplicates. The change in % HbCO will be used to calculate Hbmass. Total RBCV, PV and BV will be derived from measures of Hbmass and hematocrit29.

The collected blood samples will not be stored after the measurement.

Statistics:

A comparison of the gastric perfusion before and after chemotherapy will be performed using Friedman's test or a repeated measures ANOVA / linear mixed-effects depending on a non- or parametric nature of the data. A P-value < 0.05 will be considered significant. Statistic evaluation will be performed using IBM SPSS Statistics © (v 22.0 SPSS Inc. Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients (above 18 years) scheduled for planned open or robot-assisted resection of gastric cancer.

Exclusion Criteria:

* Allergy towards; iodine, indocyanine green or shellfish
* Severe liver insufficiency
* Thyrotoxicosis
* Nephropathy requiring dialysis
* Pregnancy or lactation
* Legally incompetent for any reason
* Withdrawal of inclusion consent
* Disseminated disease or other that contraindicates curative surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Difference in gastric perfusion | 2 years
  The primary endpoint is the difference in gastric perfusion (obtained with q-ICG, using the slope of the fluorescence curve (as described by Nerup et al)) before and after neoadjuvant chemotherapy.
  A comparison of the gastric perfusion before and after chemotherapy will be performed using Friedman's test or a repeated measures ANOVA / linear mixed-effects depending on a non- or parametric nature of the data. A P-value < 0.05 will be considered significant. Statistic evaluation will be performed using IBM SPSS Statistics © (v 22.0 SPSS Inc. Chicago, IL, USA).

SECONDARY OUTCOMES:
Short term outcome | 30 days after surgery
  postoperative events and complications as graded by the Dindo-Clavien classification
Short term outcome | 30 days after surgery
  Postoperative events as graded by the Comprehensive Complication Index
Short term outcome | 30 days after surgery
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jens TF Osterkamp, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, KBH Ø, Denmark

REFERENCES:
- [Background] Simonsen C, de Heer P, Bjerre ED, Suetta C, Hojman P, Pedersen BK, Svendsen LB, Christensen JF. Sarcopenia and Postoperative Complication Risk in Gastrointestinal Surgical Oncology: A Meta-analysis. Ann Surg. 2018 Jul;268(1):58-69. doi: 10.1097/SLA.0000000000002679. PMID 29373365
- [Background] Horowitz M, Neeman E, Sharon E, Ben-Eliyahu S. Exploiting the critical perioperative period to improve long-term cancer outcomes. Nat Rev Clin Oncol. 2015 Apr;12(4):213-26. doi: 10.1038/nrclinonc.2014.224. Epub 2015 Jan 20. PMID 25601442
- [Background] Pommergaard HC, Achiam MP, Burcharth J, Rosenberg J. Impaired blood supply in the colonic anastomosis in mice compromises healing. Int Surg. 2015 Jan;100(1):70-6. doi: 10.9738/INTSURG-D-13-00191.1. PMID 25594642
- [Background] Fawcett A, Shembekar M, Church JS, Vashisht R, Springall RG, Nott DM. Smoking, hypertension, and colonic anastomotic healing; a combined clinical and histopathological study. Gut. 1996 May;38(5):714-8. doi: 10.1136/gut.38.5.714. PMID 8707117
- [Background] Kim MJ, Shin R, Oh HK, Park JW, Jeong SY, Park JG. The impact of heavy smoking on anastomotic leakage and stricture after low anterior resection in rectal cancer patients. World J Surg. 2011 Dec;35(12):2806-10. doi: 10.1007/s00268-011-1286-1. PMID 21959931
- [Background] Kruschewski M, Rieger H, Pohlen U, Hotz HG, Buhr HJ. Risk factors for clinical anastomotic leakage and postoperative mortality in elective surgery for rectal cancer. Int J Colorectal Dis. 2007 Aug;22(8):919-27. doi: 10.1007/s00384-006-0260-0. Epub 2007 Jan 27. PMID 17260142
- [Background] Kassis ES, Kosinski AS, Ross P Jr, Koppes KE, Donahue JM, Daniel VC. Predictors of anastomotic leak after esophagectomy: an analysis of the society of thoracic surgeons general thoracic database. Ann Thorac Surg. 2013 Dec;96(6):1919-26. doi: 10.1016/j.athoracsur.2013.07.119. Epub 2013 Sep 24. PMID 24075499
- [Background] Chadi SA, Fingerhut A, Berho M, DeMeester SR, Fleshman JW, Hyman NH, Margolin DA, Martz JE, McLemore EC, Molena D, Newman MI, Rafferty JF, Safar B, Senagore AJ, Zmora O, Wexner SD. Emerging Trends in the Etiology, Prevention, and Treatment of Gastrointestinal Anastomotic Leakage. J Gastrointest Surg. 2016 Dec;20(12):2035-2051. doi: 10.1007/s11605-016-3255-3. Epub 2016 Sep 16. PMID 27638764
- [Background] Trencheva K, Morrissey KP, Wells M, Mancuso CA, Lee SW, Sonoda T, Michelassi F, Charlson ME, Milsom JW. Identifying important predictors for anastomotic leak after colon and rectal resection: prospective study on 616 patients. Ann Surg. 2013 Jan;257(1):108-13. doi: 10.1097/SLA.0b013e318262a6cd. PMID 22968068
- [Background] Thompson SK, Chang EY, Jobe BA. Clinical review: Healing in gastrointestinal anastomoses, part I. Microsurgery. 2006;26(3):131-6. doi: 10.1002/micr.20197. PMID 16518804
- [Background] Christensen JF, Jones LW, Tolver A, Jorgensen LW, Andersen JL, Adamsen L, Hojman P, Nielsen RH, Rorth M, Daugaard G. Safety and efficacy of resistance training in germ cell cancer patients undergoing chemotherapy: a randomized controlled trial. Br J Cancer. 2014 Jul 8;111(1):8-16. doi: 10.1038/bjc.2014.273. Epub 2014 May 27. PMID 24867693
- [Background] Garski TR, Staller BJ, Hepner G, Banka VS, Finney RA Jr. Adverse reactions after administration of indocyanine green. JAMA. 1978 Aug 18;240(7):635. doi: 10.1001/jama.240.7.635b. No abstract available. PMID 671679
- [Background] Alander JT, Kaartinen I, Laakso A, Patila T, Spillmann T, Tuchin VV, Venermo M, Valisuo P. A review of indocyanine green fluorescent imaging in surgery. Int J Biomed Imaging. 2012;2012:940585. doi: 10.1155/2012/940585. Epub 2012 Apr 22. PMID 22577366
- [Background] Baiocchi GL, Diana M, Boni L. Indocyanine green-based fluorescence imaging in visceral and hepatobiliary and pancreatic surgery: State of the art and future directions. World J Gastroenterol. 2018 Jul 21;24(27):2921-2930. doi: 10.3748/wjg.v24.i27.2921. PMID 30038461
- [Background] Mangano A, Fernandes E, Gheza F, Bustos R, Chen LL, Masrur M, Giulianotti PC. Near-Infrared Indocyanine Green-Enhanced Fluorescence and Evaluation of the Bowel Microperfusion During Robotic Colorectal Surgery: a Retrospective Original Paper. Surg Technol Int. 2019 May 15;34:93-100. PMID 30716160
- [Background] Zehetner J, DeMeester SR, Alicuben ET, Oh DS, Lipham JC, Hagen JA, DeMeester TR. Intraoperative Assessment of Perfusion of the Gastric Graft and Correlation With Anastomotic Leaks After Esophagectomy. Ann Surg. 2015 Jul;262(1):74-8. doi: 10.1097/SLA.0000000000000811. PMID 25029436
- [Background] Mangano A, Gheza F, Chen LL, Minerva EM, Giulianotti PC. Indocyanine Green (Icg)-Enhanced Fluorescence for Intraoperative Assessment of Bowel Microperfusion During Laparoscopic and Robotic Colorectal Surgery: The Quest for Evidence-Based Results. Surg Technol Int. 2018 Jun 1;32:101-104. PMID 29611153
- [Background] Gossedge G, Vallance A, Jayne D. Diverse applications for near infra-red intraoperative imaging. Colorectal Dis. 2015 Oct;17 Suppl 3:7-11. doi: 10.1111/codi.13023. PMID 26394736
- [Background] Watanabe J, Ishibe A, Suwa Y, Suwa H, Ota M, Kunisaki C, Endo I. Indocyanine green fluorescence imaging to reduce the risk of anastomotic leakage in laparoscopic low anterior resection for rectal cancer: a propensity score-matched cohort study. Surg Endosc. 2020 Jan;34(1):202-208. doi: 10.1007/s00464-019-06751-9. Epub 2019 Mar 14. PMID 30877565
- [Background] Sujatha-Bhaskar S, Jafari MD, Stamos MJ. The Role of Fluorescent Angiography in Anastomotic Leaks. Surg Technol Int. 2017 Jul 25;30:83-88. PMID 28277591
- [Background] Alekseev M, Rybakov E, Shelygin Y, Chernyshov S, Zarodnyuk I. A study investigating the perfusion of colorectal anastomoses using fluorescence angiography: results of the FLAG randomized trial. Colorectal Dis. 2020 Sep;22(9):1147-1153. doi: 10.1111/codi.15037. Epub 2020 Apr 6. PMID 32189424
- [Background] Ladak F, Dang JT, Switzer N, Mocanu V, Tian C, Birch D, Turner SR, Karmali S. Indocyanine green for the prevention of anastomotic leaks following esophagectomy: a meta-analysis. Surg Endosc. 2019 Feb;33(2):384-394. doi: 10.1007/s00464-018-6503-7. Epub 2018 Nov 1. PMID 30386983
- [Background] Nerup N, Andersen HS, Ambrus R, Strandby RB, Svendsen MBS, Madsen MH, Svendsen LB, Achiam MP. Quantification of fluorescence angiography in a porcine model. Langenbecks Arch Surg. 2017 Jun;402(4):655-662. doi: 10.1007/s00423-016-1531-z. Epub 2016 Nov 15. PMID 27848028
- [Background] Bell ML, Kenward MG, Fairclough DL, Horton NJ. Differential dropout and bias in randomised controlled trials: when it matters and when it may not. BMJ. 2013 Jan 21;346:e8668. doi: 10.1136/bmj.e8668. PMID 23338004
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Owens SL. Indocyanine green angiography. Br J Ophthalmol. 1996 Mar;80(3):263-6. doi: 10.1136/bjo.80.3.263. No abstract available. PMID 8703866
- [Background] Spinoglio G, Bertani E, Borin S, Piccioli A, Petz W. Green indocyanine fluorescence in robotic abdominal surgery. Updates Surg. 2018 Sep;70(3):375-379. doi: 10.1007/s13304-018-0585-6. Epub 2018 Aug 29. PMID 30159820

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT05354856/Prot_SAP_000.pdf